CLINICAL TRIAL: NCT06746701
Title: Investigating the Clinical Cure Rate and the Risk Reduction of Hepatocellular Carcinoma in Chronic HBV Infected Individuals With a Family History of Liver Cancer Using PegIFN α-2b Combined With NA Treatment in a Real-world Study.
Brief Title: Study on the Treatment of Hepatitis B Virus(HBV) Infected Individuals With Peginterferon α-2b Combined With NA.
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202207428
Record Dates: First submitted 2024-12-10; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: HBV
Keywords: Peginterferon α-2b injection; Nucleotide Analogues; HBV
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — This study is a retrospective-prospective observational study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peg-IFNα-2b combined with NA
  Interventions: Drug: Peg-IFNα-2b combined with NA
- NA monotherapy
  Interventions: Drug: Nucleotide Analogues

INTERVENTIONS:
Drug: Peg-IFNα-2b combined with NA — From baseline day 1, take NA orally once daily until the drug can be discontinued. Concurrently, combine with Peg-IFN α-2b 180μg, administered subcutaneously once a week for 48-96 weeks (if the surface antigen is not converted to negative at week 48, continue Peg-IFN α-2b treatment, but the course of treatment should not exceed 96 weeks). Discontinue Peg-IFN α-2b (while maintaining continuous oral administration of NA), and continue taking NA orally.
  Groups: Peg-IFNα-2b combined with NA
Drug: Nucleotide Analogues — Starting from the first day of enrollment, take NA orally once a day.
  Groups: NA monotherapy

SUMMARY:
This is a retrospective prospective, open-label, multicenter clinical study aiming to recruit 400 individuals with a family history of liver cancer to explore the clinical cure rate and the effectiveness, feasibility, and safety of PEGylated interferon α-2b combined with nucleos(t)ide analogues in treating chronic HBV carriers with a family history of liver cancer for reducing the risk of liver cancer occurrence. Patients will enrolled into Group A (Peg-IFNα-2b combined with NA treatment group) or Group B (NA monotherapy group) based on their medication choices. Each group is expected to enroll 200 patients, with all patients followed up to 240 weeks. The dosage, frequency, and duration of treatment with Peg-IFN α-2b and NA will be prescribed by the researchers according to clinical practice and standard treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age18-65 years (inclusive of 18 and 65), no restriction on gender;
* HBsAg positive history for at least 6 months;
* Family history of liver cancer [including first-degree and second-degree relatives; first-degree relatives are parents, children, and siblings (same parents), while second-degree relatives are uncles, aunts, grandparents, and great-grandparents; a family history of liver cancer means that one or more first-degree or second-degree relatives have had liver cancer];
* Planning to or already receiving treatment with Peginterferon alpha-2b in combination with nucleoside (acid) analogs, or receiving nucleoside (acid) analogs treatment alone;
* Negative urine or serum pregnancy test within 24 hours before the first dose (for women of childbearing age);
* Willing to receive treatment and sign an informed consent form.

Exclusion Criteria:

* Allergy to interferon;
* History of using telbivudine for antiviral treatment;
* ALT(Alanine Aminotransferase) greater than 10 times the upper limit of normal, total bilirubin greater than 2 times the upper limit of normal;
* Decompensated liver cirrhosis;
* Neutrophil count < 1.5 x 10^9/L or platelet count < 80 x 10^9/L;
* Presence of severe lesions in vital organs such as the cardiovascular, pulmonary, renal, brain, and fundus;
* Those with autoimmune diseases, psychiatric disorders, poorly controlled diabetes, or thyroid dysfunction (hyperthyroidism or hypothyroidism);
* Confirmed or suspected liver cancer or other malignant tumors;
* Post-organ transplant or preparing for organ transplantation;
* Currently using immunosuppressants;
* Pregnant or planning to become pregnant within 2 years;
* Alcohol or drug addicts;
* HIV co-infection;
* Other conditions deemed unsuitable for interferon use by the attending physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Select chronic HBV carriers with a family history of liver cancer from each center.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2029-05-25 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | through study completion, an average of 24 weeks.
  The definition of a cure is: maintaining HBsAg(Hepatitis B surface antigen) negativity (with or without the appearance of anti-HBs), undetectable HBV DNA, normal liver biochemical indices, and improvement in liver tissue lesions after discontinuation of treatment.
Liver cancer incidence rate | through study completion, an average of 24 weeks.

SECONDARY OUTCOMES:
The decrease in HBsAg compared to baseline. | through study completion, an average of 24 weeks.
HBsAg seroconversion rate | through study completion, an average of 24 weeks.
Changes of biomarkers after disease progression-related markers such as HBV DNA quantification compared to baseline. | through study completion, an average of 24 weeks.
Incidence of abnormal and clinically relevant changes in vital signs | through study completion, an average of 24 weeks.
Incidence of treatment-emergent adverse event (AE) | through study completion, an average of 24 weeks.
Incidence of abnormal and clinically relevant changes in laboratory assessments | through study completion, an average of 24 weeks.
Incidence of severe acute allergic reactions occurring during treatment. | through study completion, an average of 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: LeDu Zhou, Ph.D, Principal Investigator — Xiangya Hospital of Central South University
Locations (4):
- China (4):
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Chenzhou Second People's Hospital, Chenzhou, Hunan
  - First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Hengyang Third People's Hospital, Hengyang, Hunan

IPD SHARING:
Plan to Share IPD: No